CLINICAL TRIAL: NCT00096005
Title: A Phase I Trial Of 17-Allylaminogeldanamycin (17-AAG) And PS341 In Advanced Malignancies
Brief Title: Tanespimycin and Bortezomib in Treating Patients With Advanced Solid Tumors or Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00043; NCI-2009-00043 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0214; NCI-6121; CDR0000391837; MC0214 (Other: Mayo Clinic); 6121 (Other: CTEP); U01CA069912 (NIH); P30CA015083 (NIH); NCT01646905 (obsolete NCT alias); NCT01664325 (obsolete NCT alias)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; AIDS-related Peripheral/Systemic Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — tanespimycin; Bortezomib

ARMS (1):
- Treatment (chemotherapy and enzyme inhibitor therapy) (Experimental): Patients receive tanespimycin IV over 1-2 hours and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of tanespimycin and bortezomib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 12 additional patients are treated as above* at the MTD.
  NOTE: *Bortezomib is not administered on day 1 of course 1 only. Patients are followed at 3 months.
  Interventions: Drug: tanespimycin; Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of giving tanespimycin together with bortezomib in treating patients with advanced solid tumors or lymphomas. (Accrual for lymphoma patients closed as of 11/27/09) Drugs used in chemotherapy, such as tanespimycin, work in different ways to stop cancer cells from dividing so they stop growing or die. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. It may also increase the effectiveness of tanespimycin by making cancer cells more sensitive to the drug. Combining tanespimycin with bortezomib may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the dose-limiting toxicity and maximum tolerated dose of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) (tanespimycin) and bortezomib in patients with advanced solid tumors or lymphomas (Accrual for Lymphoma Patients Closed as of 11/27/09).

II. Determine changes in biomarkers (e.g., HSP70, client proteins, and ubiquitination of proteins) in peripheral blood mononuclear cells and tumor specimens from patients with advanced solid tumors or lymphomas (Accrual for Lymphoma Patients Closed as of 11/27/09) treated with this regimen.

III. Determine responses in patients treated with this regimen. IV. Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive tanespimycin intravenously (IV) over 1-2 hours and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of tanespimycin and bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 12 additional patients are treated as above* at the MTD.

NOTE: *Bortezomib is not administered on day 1 of course 1 only. Patients are followed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor or lymphomas (Accrual for Lymphoma Patients Closed as of 11/27/09)
* Refractory to standard treatment OR no standard treatment that is potentially curative or capable of prolonging life expectancy exists
* Tumor amenable to biopsy (patients accrued at the MTD only)
* No CNS metastases
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2 times ULN (5 times ULN if due to liver involvement)
* Creatinine ≤ 2 times ULN
* QTc < 500 msec for men (470 msec for women)
* LVEF > 40% by echocardiogram
* Ejection fraction normal by echocardiogram (for patients who have received prior anthracycline therapy)
* No cardiac symptoms ≥ grade 2
* No New York Heart Association class III or IV heart failure
* No myocardial infarction within the past year
* No active ischemic heart disease within the past year
* No congenital long QT syndrome
* No left bundle branch block
* No history of uncontrolled dysrhythmias or requiring antiarrhythmic drugs
* No history of cardiac toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine)
* No poorly controlled angina
* No history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No other significant cardiac disease
* Pulse oximetry at rest and exercise < 88% (per Medicare guidelines)
* No pulmonary symptoms ≥ grade 2
* No significant pulmonary disease requiring oxygen supplementation or causing a severe limitation in activity
* No symptomatic pulmonary disease requiring medication including any of the following:

  * Dyspnea on or off exertion
  * Paroxysmal nocturnal dyspnea
  * Oxygen requirement and significant pulmonary disease, including chronic obstructive/restrictive pulmonary disease
* No home oxygen use that meets the Medicare criteria
* No history of pulmonary toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine)
* No seizure disorder
* No sensory peripheral neuropathy > grade 1
* No neuropathic pain of any etiology

  * Patients with residual peripheral neuropathy ≤ grade 1 due to oxaliplatin therapy allowed
* No uncontrolled infection
* No prior serious allergic reaction to eggs
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to return to Mayo Clinic Rochester, Mayo Clinic Arizona, or Mayo Clinic Florida for follow up
* More than 4 weeks since prior immunotherapy or biologic therapy
* No concurrent prophylactic colony-stimulating factors
* No concurrent immunotherapy, biologic therapy, or gene therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy
* Concurrent steroids (at a stable dose for ≥ 4 weeks) for comorbid conditions (e.g., adrenal insufficiency or rheumatoid arthritis) allowed
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy that potentially included the heart in the field (e.g., mantle) or chest
* No prior radiotherapy to > 25% of bone marrow
* No prior radiopharmaceuticals
* No concurrent radiotherapy
* Recovered from prior therapy
* More than 8 weeks since prior UCN-01
* No concurrent warfarin

  * Low molecular weight heparin allowed
* No concurrent medications that prolong or may prolong QTc interval
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-11; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
MTD of tanespimycin in combination with bortezomib in the treatment of solid tumors | At 3 weeks
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of the solid tumor patients (at least 2 of a maximum of 6 new patients).
Toxicity of tanespimycin in combination with bortezomib in the treatment of solid tumors | At 3 weeks
  Defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 as adverse events that are classified as either possibly, probably, or definitely related to study treatment. Non-hematologic toxicities will be evaluated via the ordinal common toxicity criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading.
Changes in biomarkers in peripheral blood mononuclear cells and tumor specimens from patients with advanced solid tumors or lymphomas | Baseline, days 4, 8, and 11 of course 1, and at the end of treatment study
  Changes in the levels of expressions of HSP70, client proteins, and ubquitination of proteins in PBMC at the different dose levels as well as at the different time points will be descriptively summarized. The degree of proteasome inhibition will be quantitated whenever possible and the results will be displayed graphically and analyzed using simple descriptive statistics.
Responses in patients treated with this regimen | Every 6 weeks
  Evaluated using the modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease (overall and by tumor group).
Time until hematologic nadirs (WBC, ANC, platelets) | Days 4, 8, and 11 of course 1 and then every 21 days
Time to progression | Every 6 weeks
Time to treatment failure | At 3 weeks and every 6 weeks
  Defined as the time from registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States